CLINICAL TRIAL: NCT02257996
Title: The Effectiveness of Online Systematic Brief Psychodynamic Psychotherapy Via HIPAA Complaint Web Conferencing on Adults With Neurotic Disorders: a Randomized Controlled Trial
Brief Title: Effectiveness of Online Systematic Brief Psychodynamic Psychotherapy for Neurotic Disorders: Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Claudia Catao Alves Siqueira, PhD researcher, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBPP-1
Record Dates: First submitted 2014-09-24; First posted 2014-10-07 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Neurotic Disorders
Keywords: Psychoanalytic Psychotherapy; Telepsychology; Online Therapy; Web conferencing; RCT; HIPAA
MeSH Terms: conditions — Neurotic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional Group (Experimental): Online Systematic Brief Psychodynamic Psychotherapy
  Interventions: Behavioral: Online Systematic Brief Psychodynamic Psychotherapy
- Control Group (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: Online Systematic Brief Psychodynamic Psychotherapy — Systematic Adaptative Diagnosis System will be applied in both groups at two different times: pre-treatment and post-treatment
  Arms: Interventional Group

SUMMARY:
Objective: To evaluate the effectiveness of online systematic brief psychodynamic psychotherapy (SBPP) via HIPAA compliant web conferencing on adults with neurotic disorders.

Design: Randomized controlled trial. Single blind.

Setting: Internet users in the community, in São Paulo, Brazil.

Participants: Thirty-two adults will be randomly allocated to a group will receive online systematic brief psychodynamic psychotherapy (n=16), or a waiting list group (n=16).

Method: Systematic adaptative diagnosis system will be applied in both groups at pre-treatment and post-treatment (or post-waiting list). Assessment will be a comparison of the adaptative diagnosis evolution between groups.

Primary Outcomes: The subjects treated with online brief systematic psychodynamic psychotherapy will present an increase in their adaptative efficacy measured by systematic adaptative diagnosis scale (SADS) in comparison to the waiting list group, when contrasting their initial and final adaptative diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Residents in Sao Paulo city,
* Graduation complete or in course,
* Fluent Portuguese,
* Basic skills on english language,
* If in psychiatric treatment, must be under treatment with stable dosage of psychiatric medication for at least 6 months,
* Participants with diagnosis of neurotic disorders (F03.650),
* Motivation for the therapeutic process,
* Availability for 4 months of psychotherapy,
* A personal computer (with an IP address), a web camera, a microphone, access to a 1 Mbps internet connection and specific computer configuration to access the Secure Psychotherapy Virtual Environment,
* Basic knowledge of elementary internet tools,
* A justified reason that impedes a in person psychotherapy, such as the ones below:

  * Lack of financial resources,
  * Frequent change of address due to work reasons,
  * Mobility restrictions related to accidents, illnesses or physical deficiencies,
  * Inability to arrive for psychotherapy appointments due to urban chaos.

Exclusion Criteria:

Participants that present:

* a schizophrenia diagnostic or any other severe mental illness,
* drug and alcohol dependence that are in abstinence from substance abuse,
* untreated diagnosis of illnesses that may cause emotional imbalance, such as thyroid malfunction,
* Participants that are undergoing a therapeutic process during the time of the research,
* Individuals with both suicidal ideation and clear intent and need emergency treatment,
* Participants do not possess the characteristics needed to be included in the sample or are bearers of deficiencies that may compromise the treatment mediated by a computer.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-05 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change in Systematic Adaptive Diagnosis Scale (SADS) | Each participant will be followed, an expected average of 3 months.
  Participants of interventional group will be followed for the duration of therapeutic process, an expected average of 3 months.
  Participants of control group will be followed after waiting-list period, an expected average of 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia CA Siqueira, MSc, Principal Investigator — University of Sao Paulo
Locations (1):
- Clinical Psychology Department from Institute of Psychology at University of Sao Paulo, São Paulo, São Paulo, Brazil